CLINICAL TRIAL: NCT05529134
Title: A Double-blind, Randomized, Intra-patient Placebo- Controlled, Multiple Dose Study of PTW-002 Evaluating Safety, Proof of Mechanism, Preliminary Efficacy, and Systemic Exposure in Patients With Dominant or Recessive Dystrophic Epidermolysis Bullosa (DDEB / RDEB) Due to Mutation(s) in Exon 73 of the COL7A1 Gene
Brief Title: Study of PTW-002 in Patients With Dominant or Recessive Dystrophic Epidermolysis Bullosa Due to Mutation(s) in Exon 73 of the COL7A1 Gene
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phoenicis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTW-002-001
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: DDEB; RDEB; exon 73; Epidermolysis Bullosa; COL7A1 gene; DEB; collagen type VII protein; C7; Dominant Dystrophic Epidermolysis Bullosa; Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTW-002 10 mg/g gel (Experimental): PTW-002 poloxamer hydrogel for topical administration (cutaneous use), 10 mg/g gel
  Interventions: Drug: PTW-002 10 mg/g gel
- Placebo (Placebo Comparator): Matching placebo poloxamer hydrogel for topical administration (cutaneous use)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTW-002 10 mg/g gel — poloxamer hydrogel for topical administration
  Arms: PTW-002 10 mg/g gel
Drug: Placebo — placebo poloxamer hydrogel for topical administration
  Arms: Placebo

SUMMARY:
A double-blind, randomized, intra-patient placebo- controlled, multiple dose study of PTW-002 evaluating safety, proof of mechanism, preliminary efficacy, and systemic exposure in patients with Dominant Dystrophic Epidermolysis Bullosa (DDEB) or Recessive Dystrophic Epidermolysis Bullosa (RDEB) due to mutation(s) in exon 73 of the COL7A1 gene. Up to two RDEB patients 4 to 17 years of age and up to 6 DDEB patients 4 years of age and older will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, and/or their legal guardian(s), if the patient is under the legal age of consent, must provide written Informed Consent or Assent, in accordance with national and/or local laws, prior to the conduct of any study related procedures. In addition, if applicable, a minor child must provide informed Assent in accordance with national and/or local laws and in compliance with the recommendations of the approving Institutional Review Board.
2. Male or female, ≥ 4 - 17 years of age at Screening for RDEB patients, and ≥ 4 years of age at Screening for DDEB patients.
3. Have a confirmed diagnosis of RDEB or DDEB and at least one pathogenic mutation in exon 73 of the COL7A1 gene. Historical genetic data may be acceptable with Medical Monitor approval.
4. Have at least one TWA that shows no signs of local infection, and contains a target lesion that is either new or has shown dynamic healing in the past and complies with the following additional criteria:

   1. surface area of the target lesion ranging from 5 to 30 cm2, located centrally in the selected TWA.
   2. exposed sub-epidermal tissue to allow absorption of the investigational medicinal product (IMP).
   3. no suspicion of current squamous cell carcinoma (SCC) upon visual inspection.
5. Have a caregiver or support person available, who can follow study instructions in compliance with the protocol and attend study site visits with the patient as required, in the opinion of the Investigator.
6. Female patients who have reached menarche and male patients must either practice true abstinence in accordance with their preferred and usual lifestyle, or agree to use acceptable, effective methods of contraception for up to 3 months following their last dose of IMP.

Exclusion Criteria:

1. Pregnant or breast-feeding female.
2. Hemoglobin level at Screening requiring transfusion. The patient may be rescreened when the condition is considered stable.
3. Use of aminoglycosides, by any route of administration, except eye drops, 7 days or 5 half-lives, whichever is longer, prior to Baseline visit.
4. Untreated carcinoma of the TWA or history of carcinoma within 5 years prior to Screening, except adequately treated cutaneous squamous or basal cell carcinoma.
5. Life expectancy less than 6 months, as assessed by the Investigator.
6. Current or known history of clinically significant hepatic or renal disease that in the opinion of the Investigator, could impact patient safety or study participation.
7. Bleeding disorder or condition, requiring the use of anticoagulants to be confirmed by activated partial thromboplastin time (aPTT) by local lab within 48 hours of first treatment.
8. Use of any investigational drug or device within 28 days or 5 half-lives of the Baseline visit, whichever is longer, or plans to participate in another study of a drug or device during the study period. The washout of 5 half-lives does not apply to gene and cell therapy.
9. History of cell therapy requiring treatment with exclusionary medication.
10. History of skin-based gene therapy to the TWA.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events (AEs)/serious adverse events (SAEs) | Baseline through Week 32
Assessment of exon 73 exclusion in COL7A1 mRNA, measured by droplet digital polymerase chain reaction (ddPCR) | Week 4

SECONDARY OUTCOMES:
Change in uptake of PTW-002 by cells at the basement membrane by fluorescent in situ hybridization (FISH) analysis | Week 4
Effect of PTW-002 on wound healing by change in wound size (surface area) | Baseline through Week 16
Effect of PTW-002 on skin strength by onset of (re)blistering of a healed wound | Baseline through Week 16
Systemic exposure through serum levels of PTW-002 after topical administration to the target wound area (TWA) | Baseline through Week 32
Effect of PTW-002 on the presence of collagen type VII protein measured by immunofluorescent staining | Week 8
Effect of PTW-002 on the presence of anchoring fibrils measured by electron microscopy | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Hal Landy, MD, Study Director — Phoenicis Therapeutics
Locations (3):
- United States (3):
  - Stanford Health Care, Stanford, California
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No